CLINICAL TRIAL: NCT03312777
Title: A Phase 1b, Double-Blind, Randomized, Placebo-Controlled, Three Segment Cross-Over Study Investigating Oral Steady-State Pharmacokinetics And Hypoalgesic Effect Of 20 Mg Omnitram And 50 Mg Tramadol In Normal Human Subjects Made Cyp2d6 Deficient By Paroxetine
Brief Title: Omnitram Pharmacokinetic and Analgesic Study Following CY2D6 Inhibition With Paroxetine In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syntrix Biosystems, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry); DF/Net Rearch (Unknown); ITT Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Omni-Pain-102
Record Dates: First submitted 2017-10-04; First posted 2017-10-18 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Pain
Keywords: analgesia, Cytochrome P450 2D6
MeSH Terms: conditions — Pain; Agnosia | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Overencapsulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Omnitram (Experimental): Oral Omnitram 20 mg (overencapsulated 10 mg tablets) administered every 6 hours for nine doses, coadministered with paroxetine.
  Interventions: Drug: Omnitram
- Tramadol (Active Comparator): Oral tramadol 50 mg (overencapsulated 50 mg tablet) administered every 6 hours for nine doses, coadministered with paroxetine.
  Interventions: Drug: Tramadol
- Placebo (Placebo Comparator): Oral placebo (overencapsulated microcrystalline) administered every 6 hours for nine doses, coadministered with paroxetine.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omnitram — Omnitram tablets overencapsulated
  Arms: Omnitram
Drug: Tramadol — Tramadol tablet overencapsulated
  Arms: Tramadol
Drug: Placebo — Microcrystalline powder overencapsulated
  Arms: Placebo

SUMMARY:
This study evaluates the analgesic effect of Omnitram and tramadol during concurrent administration of paroxetine. Paroxetine administration is expected to diminish the analgesic effect of tramadol, but not Omnitram. Each participant will receive paroxetine before and during treatment with Omnitram, tramadol, and placebo.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study to investigating the steady-state oral pharmacokinetics and hypoalgesic effects of overencapsulated: 20 mg Omnitram (2x10 mg tablets), 50 mg tramadol (1x50 mg Ultram tablet), and placebo in male and female subjects made CYP2D6 deficient by paroxetine coadministration.

Sixty participants in normal health, 18 to 50 years of age, who meet the entry criteria, will be randomized to one of the three treatments in treatment segment 1. Each arm will ingest three consecutive 20 mg daily doses of paroxetine. Twelve hours after the first paroxetine dose, subjects will be randomized to one of the treatment sequences to ingest a total of 9 doses of Omnitram, tramadol, or placebo (one dose every 6 hours). Immediately before the 9th dose a blood sample will be collected to quantify plasma Omnitram, tramadol, and paroxetine. After the 9th study drug dose, six blood samples will be collected (1.0, 1.5, 2.0, 2.5, 4.0, and 8.0 hours after the 9th dose is administered) to quantify the Omnitram and tramadol. After the 9th dose, pain tolerance will be assessed with a cold pressor test (immersion of hand in ice cold water). Participants will washout for 11-15 days after treatment 1 and treatment 2. The study will analyze treatment side effects, the pharmacokinetics, and pain tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females with normal vital signs: systolic blood pressure > 90 mm Hg and < 140 mm Hg; diastolic blood pressure > 45 mm Hg and < 90 mm Hg; pulse 40 to 100 beats per minute; respiratory rate 10 to 20 breathes per minute.
2. Between the ages of 18 and 50 years of age.
3. Able and willing to give informed consent
4. Able to comply with all study procedures.
5. If female, must not be of childbearing potential or must agree to use one or more of the following forms of contraception during screening and for 30 days following study drug administration: hormonal (e.g., oral, transdermal, intravaginal, implant or injection); double barrier (i.e., condom, diaphragm with spermicide); intrauterine device (IUD) or system (IUS); vasectomized partner (6 months minimum); abstinence; or bilateral tubal ligation.
6. Have adequate hematologic function as evidenced by the following screening results:

   WBC >3,500/mm3 and < 12,000/mm3 Platelet Count > 150,000/mm3 and < 540,000/mm3 Hemoglobin > 12.0 gm/dL and < 20.5 gm/dL

   Have adequate liver function as evidenced by the following screening results:

   AST (SGOT) ≤ 60 IU/L ALT (SGPT) men ≤ 83 IU/L women < 60 IU/L Alkaline Phosphatase ≤ 200 IU/L Total Bilirubin ≤ 1.2 mg/dL PT and PTT < 1.2 ULN
7. Electrocardiogram (ECG) without clinically significant findings as determined by the PI.
8. Have adequate renal function as evidenced by the following screening result:

   Glomerular filtration rate (GFR) calculated by Cockcroft-Gault formula >60 ml/min.

   Urinalysis demonstrating < +1 glucose, +1 ketones, and +1 protein.
9. Negative pregnancy test within 1 week of study day 1 (women of childbearing potential only).
10. Negative urine test for substances of abuse, including opiates, per CRU standards.
11. Negative serology tests for HIV, hepatitis B surface antigen, and hepatitis C virus antibody.
12. Body Mass Index (BMI) 18.0 to 32 kg/m.
13. Cold pressor screening results as follows: 1) pain tolerance of > 20 seconds and <120 seconds.
14. Cytochrome P450 2D6 (CYP2D6) genotype by Genelex consistent with intermediate metabolizer phenotype or normal metabolizer phenotype.

Exclusion Criteria:

1. Oral temperature > 38°C or history of current illness.
2. History of seizures, epilepsy, or recognized increase risk of seizure (e.g., head trauma, metabolic disorders, alcohol or drug withdrawal).
3. History of cirrhosis or laboratory evidence of liver disease.
4. Use of alcohol within 24 hours of day -1 until the end of the study; and grapefruit, grapefruit-related citrus fruits (e.g., Seville oranges, pomelos), or grapefruit juice or grapefruit-related juices, or other medication, within 7 days of study drug administration and until the end of the study.
5. History of previous anaphylaxis, severe allergic reaction to paroxetine, tramadol, codeine, or other opioid drugs.
6. Use of MAO Inhibitors (including linezolid), Serotonin Reuptake Inhibitors, Serotonin-Norepinephrine Reuptake Inhibitors, and prescription or over-the counter (OTC) medications known to induce or inhibit drug metabolism, including CYP2D6, and other drugs that may affect the serotonergic neurotransmitter systems including, but not limited to, triptans, dextromethorphan, tricyclic antidepressants, bupropion, lithium, tramadol, dietary supplements such as tryptophan and St. John's Wort, and antipsychotics or other dopamine antagonists. These restrictions are to be maintained from 14 days before study day -1, until the subject completes the study.
7. Any other unstable acute or chronic disease that could interfere with the evaluation of the safety of the study drug as determined by the principal Investigator in dialogue with the Sponsor Medical Monitor.
8. Currently pregnant or breast feeding.
9. Unlikely to comply with the study protocol.
10. Known or suspected alcohol or drug abuse within the past 6 months.
11. Received another investigational agent within 4 weeks of Day 1, or receiving any other investigational agent during this study.
12. Any concurrent disease or condition that in the opinion of the investigator impairs the subject's ability to complete the trial. Psychological, familial, sociological, geographical or medical conditions which, in the Investigator's opinion, could compromise compliance with the objectives and procedures of this protocol, or obscure interpretation of the trial data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-22 (Actual)

PRIMARY OUTCOMES:
Cold Pressor Test - Cold Water Induced-Pain | The test is performed on Day 3, shortly after the ninth (final) dose of study drug.
  The participant immerses a hand in cold water for a maximum of 3 minutes and reports the pain they experience using a "0 (no pain) to 10 (worst pain)" scale. Immersion of hand in ice cold water

SECONDARY OUTCOMES:
Adverse Events | Participant report adverse events throughout study enrolment; investigators observe adverse events during all three 3 day inpatient treatment segments; laboratory safety labs are obtained on Day 3 of treatment segment 3 (the final treatment segment).
  Adverse events will include: 1) reports by participants; 2) observations by investigators; and 3) abnormal laboratory safety test results.
Steady State Pharmacokinetics | 8 hours
  Study drug plasma concentrations are assessed using specimens collected immediately before and after the 9th dose of each treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn L Searle, MD, Principal Investigator — PRA Health Sciences; Stuart Kahn, MD, Study Director — Syntrix Biosystems
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zebala JA, Searle SL, Webster LR, Johnson MS, Schuler AD, Maeda DY, Kahn SJ. Desmetramadol Has the Safety and Analgesic Profile of Tramadol Without Its Metabolic Liabilities: Consecutive Randomized, Double-Blind, Placebo- and Active Comparator-Controlled Trials. J Pain. 2019 Oct;20(10):1218-1235. doi: 10.1016/j.jpain.2019.04.005. Epub 2019 Apr 18. PMID 31005596